CLINICAL TRIAL: NCT06233500
Title: Macular Micro Vascular Changes Following Macular Hole Repair : Optical Coherence Tomography Angiography Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fayoum University (Other)
Collaborators: Research Institute of Ophthalmology, Egypt (Other)
Responsible Party: Principal Investigator, Mohamed Hussein, Dr., Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FayoumU_28
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Macular Holes
Keywords: macular hole; ILM peeling; Temporal flap; OCTA; Optical Coherence Tomography Angiography
MeSH Terms: conditions — Retinal Perforations | interventions — Predictive Value of Tests

STUDY DESIGN:
Intervention Model Description: This study will include 28 eyes with idiopathic full thickness macular hole; All eyes in this study will be subjected to pars plana vitrectomy procedure, they will be divided into two groups:
  Group A: 16 eyes will be treated with only wide internal limiting membrane (ILM) peeling up to the arcades without ILM flap Group B : 16 eyes will be treated by ILM peeling with ILM flap.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: eyes will be treated without ILM flap (Active Comparator): Group A: Only wide ILM peeling up to the arcades well be done
  Interventions: Procedure: pars plana vitrectomy
- Group B : eyes will be treated by ILM flap (Active Comparator): Group B: ILM peeling with flap well be done
  Interventions: Procedure: pars plana vitrectomy

INTERVENTIONS:
Procedure: pars plana vitrectomy — All eyes in this study will be subjected to pars plana vitrectomy procedure with these main steps:
  * 23 G trocar system will be used
  * Posterior vitreous detachment will be induced with the aid of triamcinolone acetate injection, and core vitrectomy will be done
  * Brilliant blue stain will be injected, and ILM forceps will be used for ILM peeling
  Patients will be divided then into two groups:
  Group A: Only wide ILM peeling up to the arcades well be done Group B: ILM peeling with flap well be done
  * Shaving of the vitreous base, and then fluid air exchange
  * SF 6 gas tamponade will be used
  Other Names: PPV with ILM peeling

SUMMARY:
The goal of this prospective interventional study is to to compare the micro vascular and structural changes between surgery with and without ILM flap to repair macular hole.

The main questions it aims to answer are:

* What are the macular micro vascular and structural changes pre and post repair of idiopathic full thickness macular hole and what is the correlation between these changes and visual recovery.
* Is there are any prognostic values of the micro vascular status of the macula could be assessed preoperatively.
* What are the differences regarding these micro vascular and structural changes between repair with and without ILM flap.

Participants will be:

* Subjected to pars plana vitrectomy to repair macular hole.
* Examined by optical coherence tomography angiography pre and post operative

Researchers will compare:

Group A: eyes treated without ILM flap Group B : eyes treated by ILM flap to see if there are differences regarding the micro vascular and structural changes in the macular area.

DETAILED DESCRIPTION:
This study will include 28 eyes with idiopathic full thickness macular hole; they will be divided into two groups:

Group A: 14 eyes will be treated without ILM flap Group B : 14 eyes will be treated by ILM flap

* Sample size: 28 eyes. (based on ELM recovery rate in ILM flap 70% versus 21.4% with inverted flap (Iwasaki et al., 2019), and at power of study 80% and confidence level 95%, sample size is calculated using openEpi software to be 14 eyes in each group
* Study setting: Ophthalmology Department, Fayoum University and the Research Institute of Ophthalmology
* Data Collection :

  * History :

    1. Demographic data ( age , gender )
    2. General medical history ( DM, HTN )
    3. Symptom duration
    4. Previous ocular history
  * Clinical examination:

    1. Best corrected visual acuity using snellen chart (converted to log MAR for statiscal analysis).
    2. Slit lamp biomicroscopy for anterior segment examination.
    3. Posterior segment examination using binocular indirect ophthalmoscope and indirect slit lamp bio microscopy (+90 volk lens for detailed evaluation of macula)
    4. Axial length measurement
  * Optical Coherence Tomography:

We use SD- OCT and OCTA for pre and post-operative evaluation of retinal layers microstructure and vasculature.

* Surgical Procedure

All eyes in this study will be subjected to pars plana vitrectomy procedure with these main steps:

* 23 G trocar system will be used
* Posterior vitreous detachment will be induced with the aid of triamcinolone acetate injection, and core vitrectomy will be done
* Brilliant blue stain will be injected, and ILM forceps will be used for ILM peeling

Patients will be divided then into two groups:

Group A: Only wide ILM peeling up to the arcades well be done Group B: ILM peeling with flap well be done

* Shaving of the vitreous base, and then fluid air exchange
* SF 6 gas tamponade will be used

  • Study procedures:

  o Regular clinical assessment pre and at 1 and 6 months post-operative including:
* Best corrected visual acuity measurement using Snellen chart with conversion to log. MAR notation for statistical analysis
* Posterior segment examination using binocular indirect ophthalmoscope and indirect slit lamp bio microscopy (+90 volk lens for detailed evaluation of macula)

  * Standard Optical coherence tomography of the macula at 1 and 6 months post-operative using (SD-OCT) scans (512 A-scans, 20°×20°) with the following protocol:

Macula thickness map for measurement of central retinal thickness, and photoreceptor inner segment/outer segment complex.

o Optical coherence tomography angiography of the macula at 1 and 6 months post-operative studying Superficial Capillary plexus, Deep Capillary plexus and Fovea avascular zone.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic full thickness Macular hole without retinal detachment

Exclusion Criteria:

* Previous pars plana vitrectomy
* High myopia with axial length ≥ 26 mm.
* Uncertain symptom duration or ≥ 6 month .
* History of same eye trauma
* Poor image quality.
* Patients with diabetic retinopathy or other retinal diseases, e.g. ischemic, inflammatory.
* Any patient with significant cataract which needs combined phaco-vitrectomy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
visual acuity | It will be measured preoperative and at 1 and 6 months post-operative
  Best corrected visual acuity measurement using Snellen chart with conversion to log. MAR notation for statistical analysis
Fovea avascular zone FAZ | It will be measured preoperative and at 1 and 6 months post-operative
  Optical coherence tomography angiography used to measure FAZ area in mm2 (mm square)

SECONDARY OUTCOMES:
central retinal thickness | It will be measured preoperative and at 1 and 6 months post-operative
  Standard Optical coherence tomography of the macula using (SD-OCT) scans (512 A-scans, 20°×20°) to measure central retinal thickness in µm

CONTACTS AND LOCATIONS:
Overall Officials: Islam Mohalhal, MD, Study Director — Research Institute of Ophthalmology, Egypt
Locations (1):
- research institute of ophthalmology, Egypt, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: data will become available before the end of 2024 and will be available for 1 year
Access Criteria: it will be shared via E-mail

REFERENCES:
- [Background] Demirel S, Degirmenci MFK, Bilici S, Yanik O, Batioglu F, Ozmert E, Alp N. The Recovery of Microvascular Status Evaluated by Optical Coherence Tomography Angiography in Patients after Successful Macular Hole Surgery. Ophthalmic Res. 2018;59(1):53-57. doi: 10.1159/000484092. Epub 2017 Nov 29. PMID 29183023
- [Background] Kelly NE, Wendel RT. Vitreous surgery for idiopathic macular holes. Results of a pilot study. Arch Ophthalmol. 1991 May;109(5):654-9. doi: 10.1001/archopht.1991.01080050068031. PMID 2025167
- [Background] Lai MM, Williams GA. Anatomical and visual outcomes of idiopathic macular hole surgery with internal limiting membrane removal using low-concentration indocyanine green. Retina. 2007 Apr-May;27(4):477-82. doi: 10.1097/01.iae.0000247166.11120.21. PMID 17420702
- [Background] Casini G, Mura M, Figus M, Loiudice P, Peiretti E, De Cilla S, Fuentes T, Nasini F. INVERTED INTERNAL LIMITING MEMBRANE FLAP TECHNIQUE FOR MACULAR HOLE SURGERY WITHOUT EXTRA MANIPULATION OF THE FLAP. Retina. 2017 Nov;37(11):2138-2144. doi: 10.1097/IAE.0000000000001470. PMID 28129215
- [Background] Yun C, Ahn J, Kim M, Kim JT, Hwang SY, Kim SW, Oh J. Characteristics of retinal vessels in surgically closed macular hole: an optical coherence tomography angiography study. Graefes Arch Clin Exp Ophthalmol. 2017 Oct;255(10):1923-1934. doi: 10.1007/s00417-017-3742-6. Epub 2017 Jul 25. PMID 28744658
- [Background] Woon WH, Greig D, Savage MD, Wilson MC, Grant CA, Mokete B, Bishop F. Movement of the inner retina complex during the development of primary full-thickness macular holes: implications for hypotheses of pathogenesis. Graefes Arch Clin Exp Ophthalmol. 2015 Dec;253(12):2103-9. doi: 10.1007/s00417-015-2951-0. Epub 2015 Feb 13. PMID 25673252
- [Background] Itoh Y, Inoue M, Rii T, Ando Y, Hirakata A. Asymmetrical recovery of cone outer segment tips line and foveal displacement after successful macular hole surgery. Invest Ophthalmol Vis Sci. 2014 May 6;55(5):3003-11. doi: 10.1167/iovs.14-13973. PMID 24736052
- [Background] Spaide RF, Klancnik JM Jr, Cooney MJ. Retinal vascular layers imaged by fluorescein angiography and optical coherence tomography angiography. JAMA Ophthalmol. 2015 Jan;133(1):45-50. doi: 10.1001/jamaophthalmol.2014.3616. PMID 25317632
- [Background] Lupidi M, Coscas F, Cagini C, Fiore T, Spaccini E, Fruttini D, Coscas G. Automated Quantitative Analysis of Retinal Microvasculature in Normal Eyes on Optical Coherence Tomography Angiography. Am J Ophthalmol. 2016 Sep;169:9-23. doi: 10.1016/j.ajo.2016.06.008. Epub 2016 Jun 11. PMID 27296485
- [Background] Samara WA, Say EA, Khoo CT, Higgins TP, Magrath G, Ferenczy S, Shields CL. CORRELATION OF FOVEAL AVASCULAR ZONE SIZE WITH FOVEAL MORPHOLOGY IN NORMAL EYES USING OPTICAL COHERENCE TOMOGRAPHY ANGIOGRAPHY. Retina. 2015 Nov;35(11):2188-95. doi: 10.1097/IAE.0000000000000847. PMID 26469536
- [Background] Kim YJ, Jo J, Lee JY, Yoon YH, Kim JG. Macular capillary plexuses after macular hole surgery: an optical coherence tomography angiography study. Br J Ophthalmol. 2018 Jul;102(7):966-970. doi: 10.1136/bjophthalmol-2017-311132. Epub 2017 Oct 5. PMID 28982954